CLINICAL TRIAL: NCT03075059
Title: Child Life Intervention to Decrease Anxiety in Patients and Caregivers for Outpatient Surgical Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Marleta Reynolds, MD, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-161
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Surgery
MeSH Terms: interventions — Allied Health Personnel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): For patients randomized to the intervention group, the Child Life specialist will reach out via telephone to offer support and expertise in helping prepare their child and themselves for outpatient surgery to help decrease anxiety and increase coping. Concepts covered will include: developmentally appropriate language for explaining surgery and related procedures, potential coping skills to ease separation for caregivers and pediatric patients. Additionally, written materials (attached) covering the same information will be sent via mail or email covering the same information discussed in the phone conversation to serve as a refresher and resource before the day of surgery. On the day of surgery, the patient will receive standard of care (SOC) Child Life Services available to all patients.
  Interventions: Behavioral: Child Life
- Control (No Intervention): Patients randomized to the control group will not receive the preoperative phone call or written materials and will only receive SOC Child Life services on the day of surgery.

INTERVENTIONS:
Behavioral: Child Life — For patients randomized to the intervention group, the Child Life specialist will reach out via telephone to offer support and expertise in helping prepare their child and themselves for outpatient surgery to help decrease anxiety and increase coping. Concepts covered will include: developmentally appropriate language for explaining surgery and related procedures, potential coping skills to ease separation for caregivers and pediatric patients. Additionally, written materials (attached) covering the same information will be sent via mail or email covering the same information discussed in the phone conversation to serve as a refresher and resource before the day of surgery. On the day of surgery, the patient will receive standard of care (SOC) Child Life Services available to all patients.
  Arms: Intervention

SUMMARY:
1. Determine preoperative and postoperative levels of anxiety for pediatric patients ages 6-17 related to outpatient surgical intervention using the validated Psychosocial Risk Assessment in Pediatrics (PRAP) assessment tool, the State-Trait Anxiety Inventory for Adults(STAI-AD), and the State-Trait Anxiety Inventory for Children (STAI-CH)
2. Determine preoperative and postoperative levels of anxiety for parent/guardian of pediatric patients ages 6 - 17 related to outpatient surgical intervention using the validate PsychosocialRisk Assessment in Pediatrics (PRAP) assessment tool and the State-Trait Anxiety Inventory for Adults (STAI-AD).
3. Assess if additional Child Life intervention offered pre-operatively to one group demonstrates differences in PRAP scores compared to control group

DETAILED DESCRIPTION:
This is a prospective, interventional study with two groups of patients scheduled for outpatient surgery at Ann and Robert H. Lurie Children's Hospital of Chicago. Participants eligible for enrollment will be identified and screened upon diagnosis and/or at the time of referral for surgery until patient enrollment is completed. Based on a power analysis, using average scores and norms for the validated tool with a projected difference of four points difference between groups, minimum enrollment is 22 per group, 44 patients total to detect a statistically significant difference based on established parameters.

Potential participants will be identified in the outpatient clinic setting once a physician and family has agreed to pursue surgical invention. The research team will consent either during clinical evaluation or following surgical consent obtainment. All questions will be answered prior to obtaining signed study consent. Once consent is received, Child Life will be paged to observe the patient and caregiver along with the physician provider in order to observe and assess behavior required to complete the PRAP assessment form. Additionally, the patient and parent/guardian will be asked to complete the STAI-CH and STAI-AD assessments as appropriate per age. After the completion of the assessments the patient and family will be randomly assigned to intervention or control group. Only the Child Life Specialist and research staff facilitating the intervention will be unblinded as to which patients are in which group, which is necessary for conducting the study. All other study staff will remain blinded. For patients randomized to the intervention group, the Child Life specialist will reach out via telephone to offer support and expertise in helping prepare their child and themselves for outpatient surgery to help decrease anxiety and increase coping. Concepts covered will include: developmentally appropriate language for explaining surgery and related procedures, potential coping skills to ease separation for caregivers and pediatric patients. Additionally, written materials (attached) covering the same information will be sent via mail or email covering the same information discussed in the phone conversation to serve as a refresher and resource before the day of surgery. On the day of surgery, the patient will receive standard of care (SOC) Child Life Services available to all patients. Patients randomized to the control group will not receive the preoperative phone call or written materials and will only receive SOC Child Life services on the day of surgery.

After the surgical induction or day of the procedure, the Child Life Specialist will complete the PRAP and document in EPIC per SOC procedures. The Child Life Specialist will also attend the postoperative and complete the third PRAP based on feedback from the patient, family/caregiver and providing surgeon. At this postoperative time the patient and parent/guardian will be asked to complete the STAI-CH and STAI-AD assessments as appropriate per age for the second time. Once data is collected, analysis will compare PRAP, STAI-CH, and STAI-AD scores between groups at all three points on the timeline. Information gained may be used to help direct and develop interventions to help decrease patient and family anxiety and increase coping related to surgical intervention

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients ages 6 - 17 and their families/caregivers that are scheduled for outpatient surgical intervention in the division of pediatric surgery of Ann and Robert H. Lurie Children's Hospital of Chicago. Patients receiving low acute, lower risk procedures will be enrolled

Exclusion Criteria:

* Patients who may turn 18 during the course of the study will not be eligible for enrollment and will be excluded.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient and Parent/Guardian State and Trait Anxiety | 6 months
  Patient and Parent/Guardian State and Trait Anxiety is measured using the the State-Trait Anxiety Inventory for Adults (STAI-AD), and the State-Trait Anxiety Inventory for Children (STAI-CH) for children between the ages of 6 and 14

SECONDARY OUTCOMES:
Patient and Parent/Guardian PRAP scores | 6 months
  Patient and Parent/Guardian Anxiety is also measured using the Psychosocial Risk Assessment in Pediatrics (PRAP) assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Marleta Reynolds, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No